CLINICAL TRIAL: NCT07150078
Title: Investigation of Differences in Dual and Single Motor and Cognitive Tasks of Children With Attention Deficit and Hyperactivity Disorder Compared to Healthy Children
Brief Title: Dual Task and Attention Deficit and Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Zekiye İpek, Assoc.Prof, Gaziantep Islam Science and Technology University
Other Study IDs: ipekkirmaci.
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: dual task; motor performance; cognitive perfomance
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD: Attention Deficit Hyperactivity Disorder (ADHD): All tests will be applied to ADHD children.
  Interventions: Diagnostic Test: test
- Control: Healthy Children: All tests will be applied to healthy children.
  Interventions: Diagnostic Test: test

INTERVENTIONS:
Diagnostic Test: test — Descriptive tests will be applied

SUMMARY:
When motor control deficits, sensory-perceptual deficits, and deficits in attention allocation and executive functions, often seen in ADHD, are accompanied by impairments in attentional allocation and executive function, further difficulties with dual tasks may arise. The aim of this study was to compare the performance of children diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) with healthy children on single-motor and dual-motor and motor-cognitive tasks.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD), characterized by inattention, hyperactivity, and impulsivity, is a heterogeneous neurodevelopmental disorder frequently encountered in childhood. Genetic, social, and physical factors play a significant role in ADHD, and it is known that it can cause problems in many areas, including financial costs, family responsibilities, academic performance, and physical and mental health. These children are fidgety, unable to sit still, boredom with sitting for long periods, constantly running or climbing in childhood, but as adults, they remain restless, often climbing walls, have difficulty engaging in quiet activities, begin speaking before the other person has even finished, interrupt others, talk excessively, and have difficulty with tasks that require waiting or taking turns. Hyperactivity is more common in these children during the preschool years. Other characteristics of these children include being stubborn, sleepy, bedwetting, and displaying anger and aggression in response to situations. Motor activity decreases with age. By adulthood, they experience emotional distress. Dual tasking, a common occurrence in daily life, is defined as the simultaneous performance of two tasks that can be performed independently, measured separately, and have different objectives. In dual tasking, motor-motor, motorcognitive, or cognitive-cognitive tasks are performed simultaneously. When motor control deficits, sensory-perceptual deficits, attention allocation, and executive function deficits frequently seen in ADHD coexist, further difficulties with dual tasks may arise.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 7 and 16,
* having been diagnosed with ADHD,
* volunteering to participate in the study, or having received parental consent.

Exclusion Criteria:

* The individual is unwilling to participate in the study or does not have family consent.
* The individual has another known neurological or orthopedic disease.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Attention Deficit and Hyperactivity Disorder and Healthy Children
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Nine hole peg test- Single task | At Baseline
  Participants are asked to place nine 3.2 cm long sticks into the holes on the platform as quickly as possible and then collect them. This process is timed and recorded in seconds.
Nine hole peg test-motor dual task | at baseline
  Participants are asked to place nine 3.2 cm long sticks into the holes on the platform as quickly as possible and then collect them. This process is timed and recorded in seconds. Keeping pace with the foot during the 9-hole peg for motor-motor dual task (dorsi-plantar flexion)
Nine hole peg test- congitive dual task | At baseline
  Participants are asked to place nine 3.2 cm long sticks into the holes on the platform as quickly as possible and then collect them. This process is timed and recorded in seconds. During the 9-hole peg test for the motor-cognitive dual task, they will be asked to say animal names starting with the letter K.
10 meter walk test-single task | at baseline
  The subject is asked to walk a 10-meter distance at a normal walking pace. To mitigate the effects of acceleration and deceleration, a 2-meter starting and finishing distance is included before and after the 10-meter test area. During the test, the timer starts when the subject's foot crosses the starting line and stops when the subject crosses the finishing line. Two measurements are taken, and the best value is recorded in m/s.
Ten meter walk test- motor dual task | At baseline
  The subject is asked to walk a 10-meter distance at a normal walking pace. To mitigate the effects of acceleration and deceleration, a 2-meter starting and finishing distance is included before and after the 10-meter test area. During the test, the timer starts when the subject's foot crosses the starting line and stops when the subject crosses the finishing line. Two measurements are taken, and the best value is recorded in m/s. For the motor-motor dual task, children will be asked to carry a tray containing an empty box with two hands during the 10-meter walking test.
Ten meter walk test- cognitive dual task | at baseline
  The subject is asked to walk a 10-meter distance at a normal walking pace. To mitigate the effects of acceleration and deceleration, a 2-meter starting and finishing distance is included before and after the 10-meter test area. During the test, the timer starts when the subject's foot crosses the starting line and stops when the subject crosses the finishing line. Two measurements are taken, and the best value is recorded in m/s. For the motor-cognitive dual task, children will be asked to say animal names starting with the letter K during the 10-meter walking test.

CONTACTS AND LOCATIONS:
Overall Officials: ipek kırmacı, Study Director — GIBTU
Locations (1):
- Ipek Kırmacı, Şehitkamil, Gaziantep, Turkey (Türkiye)